CLINICAL TRIAL: NCT07367724
Title: Safety and Efficacy of Ademetionine in Patients With Obstructive Hypertrophic Cardiomyopathy: A Multicenter, Double-Blind, Randomized Controlled, Phase 2 Study
Brief Title: Ademetionine in Obstructive Hypertrophic Cardiomyopathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-ZX068
Record Dates: First submitted 2025-12-25; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy (oHCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ademetionine group (Active Comparator)
  Interventions: Drug: Ademetionine 1,4-Butanedisulfonate
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ademetionine 1,4-Butanedisulfonate — Ademetionine 1,4-Butanedisulfonate is the currently available marketed oral pharmaceutical formulation of S-adenosylmethionine. Its brand name is Ximeixin in China.
  Arms: Ademetionine group
Drug: Placebo — The placebo is a starch tablet identical in appearance, odor, and other physical properties.
  Arms: Placebo group

SUMMARY:
This study is a multicenter, double-blind, randomized controlled Phase 2 trial designed to evaluate the safety and efficacy of Ademetionine in patients with obstructive hypertrophic cardiomyopathy (oHCM). The study will recruit patients with oHCM who, under double-blind conditions, will be randomly assigned to either the Ademetionine group or the placebo group. Follow-up visits will be conducted every 4 weeks until 16 weeks from baseline. After 16 weeks, the study will evaluating the effect of Ademetionine on exercise capacity, heart failure symptoms, cardiac structure and function, and quality of life, as well as safety and tolerability of Ademetionine in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for HCM.
* Age ≥ 18 years at screening.
* LVEF ≥ 50% at screening.
* Echocardiography demonstrates a resting or provoked LVOTG ≥ 30 mmHg at screening.
* NYHA Functional Class II-III at screening.
* Able to perform CPET, with Peak VO₂ ≤ 20 mL/kg/min at screening.
* Willing and able to sign the informed consent form and comply with all scheduled study visits.

Exclusion Criteria:

* History of severe hypersensitivity to any component of Ademetionine 1,4-Butanedisulfonate Enteric-coated Tablets.
* Known genetic defects affecting methionine cycle and/or causing homocystinuria and/or hyperhomocysteinemia (e.g., cystathionine beta-synthase deficiency, vitamin B12 metabolic defects).
* Current vitamin B12 or folate deficiency.
* History of psychiatric disorders, or current use of antidepressants such as clomipramine.
* Planned for any surgical (including septal reduction therapy) or interventional procedure during the trial period.
* Planned use of cardiac myosin inhibitors (e.g., Mavacamten) during the trial period.
* Currently pregnant or planning pregnancy.
* Currently participation in another drug or device clinical trial.
* History of any other disease with a life expectancy of less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pVO₂ by CPET from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks

SECONDARY OUTCOMES:
Proportion of participants with ≥1 class improvement in NYHA Functional Class from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks
Change in KCCQ-CSS from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks
Change in provoked left ventricular outflow tract gradient from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks
Change in left ventricular mass index from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks
Change in left atrial volume index from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks
Change in E/e' from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks
Change in VE/VCO₂ slope by CPET from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks

OTHER OUTCOMES:
Change in maximal left ventricular wall thickness from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks
  Exploratory endpoint
Change in NT-proBNP from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks
  Exploratory endpoint
Change in hs-cTnI from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks
  Exploratory endpoint
Change in hs-cTnT from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks
  Exploratory endpoint
Change in SF-36 from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks
  Exploratory endpoint
Change in HCMSQ from baseline to Week 16 | From enrollment to the end of treatment at 16 weeks
  Exploratory endpoint

IPD SHARING:
Plan to Share IPD: Undecided